CLINICAL TRIAL: NCT04444934
Title: Can Intraoperative Visual Examination of Diaphragmatic Peritoneum be a Reliable Tool to Modulate the Extent of Interval Debulking Surgery in Advanced Ovarian Cancer? The VIPER (VIsual Peritoneal Evaluation of Residual Disease) Study
Brief Title: Intra-operative Visual Examination at IDS
Acronym: VIPER
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Other Study IDs: DIPUSVSP-03-02-2033
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Diaphragm Disease
Keywords: ovarian cancer; interval debulking surgery; visual examination
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with not-surely pathologic diaphragmatic peritoneum: The definition of not-surely pathologic diaphragmatic peritoneum was given in association with the presence of flat dyschromic areas.
  Interventions: Other: histological examination
- Patients with certainly pathologic diaphragmatic peritoneum: The definition of certainly pathological diaphragmatic peritoneum was given when isolated or confluent thick nodules were visualized at the intra-operative inspection.
  Interventions: Other: histological examination

INTERVENTIONS:
Other: histological examination — Patients were classified in two groups based on the surgeon's visual examination of the right diaphragmatic peritoneum. The accuracy of visual examination has been assessed comparing surgeon's opinions to histological examination

SUMMARY:
Complete disease removal has the greatest impact in the treatment of advanced ovarian cancer, both during primary debulking surgery (PDS) and interval debulking surgery (IDS), but, contrarily to PDS, no consensus exist on the interpretation of the absence of residual tumor at IDS. In addition, chemotherapy induces fibrotic changes that can hinder the surgeon's ability to properly assess the spread of abdominal disease. The aim of the study is to evaluate the accuracy of visual inspection compared to histopathological examination at the level of the diaphragmatic peritoneum in patients undergoing surgery after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
All data of patients subjected to IDS between October 2016 and October 2019 with evidence of suspected or certain residual disease at the level of the right diaphragmatic peritoneum, at intra-operative evaluation have been collected. Diaphragmatic peritoneum was classified as negative, not-surely pathologic and certainly pathologic by the surgeon, and based on the surgeon's opinion, a diaphragmatic biopsy or peritonectomy was then performed. The definition of not-surely pathologic diaphragmatic peritoneum was given in association with the presence of flat dyschromic areas, while the definition of certainly pathological diaphragmatic peritoneum was given when isolated or confluent thick nodules were visualized at the intra-operative inspection. Residual disease was indicated at the end of each intervention and classified as no residual disease (RD=0, complete cytoreduction), less than 1 centimeter (RD </= 1 cm, optimal cytoreduction) or more than 1 cm (RD > 1 cm, sub-optimal cytoreduction).

Pathological specimens' results were also divided in negative (no evidence of disease), microscopic evidence of residual disease (</= 3 mm) or macroscopic signs of residual disease (> 3 mm). Microscopic and macroscopic disease were both considered as positive for residual disease.

General early post-operative complications (arising within 30 days from surgery), and complications related to diaphragmatic peritonectomy, as post-operative pleural effusion, were classified using the extended Clavien-Dindo classification of surgical complications.

The primary end-point of the study was to evaluate the accuracy, sensitivity and specificity of the visual inspection compared to histopathological examination, at the level of the right diaphragmatic peritoneum, in patients subjected to IDS.

The secondary endpoints were to evaluate the rate of early postoperative complications related to diaphragmatic peritonectomy and assess whether this procedure may delay the re-start of post-operative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with histology proven biopsy of epithelial ovarian, fallopian or peritoneal cancer (FIGO stage III C - IV B), judged suitable for IDS by clinicians, with evidence of suspected or certain residual disease at the level of the right diaphragmatic peritoneum, at intraoperative evaluation.

Exclusion Criteria:

* Patients with no evidence of diaphragmatic disease during IDS, and who therefore did not undergo diaphragmatic peritonectomy or biopsy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histology proven biopsy of epithelial ovarian, fallopian or peritoneal cancer (FIGO stage III C - IV B), judged suitable for IDS by clinicians, with evidence of suspected or certain residual disease at the level of the right diaphragmatic peritoneum, at intraoperative evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Accuracy | During surgery
  to evaluate the accuracy of the visual examination compared to histopathological examination, at the level of the right diaphragmatic peritoneum, in patients subjected to IDS

SECONDARY OUTCOMES:
Post-operative complications | up to 30 days after surgery
  to evaluate the rate of early postoperative complications related to diaphragmatic peritonectomy

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Costantini, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided